CLINICAL TRIAL: NCT00119665
Title: A Phase II, Double-Blind, Placebo-Controlled, Randomized Clinical Trial Assessing Toxicity and Efficacy of MF101 for Hot Flashes and Menopausal Symptoms
Brief Title: Clinical Trial Assessing Toxicity and Efficacy of MF101 for Hot Flashes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionovo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MF-101-002
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-03

CONDITIONS: Hot Flashes
Keywords: Postmenopausal symptoms; Hot Flashes; Postmenopausal Hot Flashes
MeSH Terms: conditions — Hot Flashes

INTERVENTIONS:
Drug: MF101

SUMMARY:
The researchers propose a Phase II randomized, double-blind, placebo-controlled trial of 180 healthy postmenopausal women experiencing at least 5 hot flashes per day or 35 hot flashes per week. Women will be randomized to one of three arms: 4.5 grams/day (dry weight of extract) of MF101, 9.0 grams/day (dry weight of extract) of MF101 or placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 40 to 60.
* Currently receiving medical care from a health care provider.
* Self-report 5 hot flashes per day or 35 hot flashes per week.
* Postmenopausal as defined by 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 30mlU/ml or 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy or hysterectomy with FSH levels > 30 mlU/ml.
* Agree not to start new herbal or dietary supplements and not to change the dose of any currently used herbal or dietary supplements for the duration of the trial.
* Successful completion of a Hot Flash Diary, a Daily Study Medication Diary and a Bleeding Diary, tolerates placebo, and 80% compliant at run-in.
* Must have had a mammogram within the last 9 months.
* Have access to a phone.
* Provide informed consent.

Exclusion Criteria:

* Inability to sign an informed consent or fill out questionnaires.
* History of breast, uterine or ovarian cancer or melanoma.
* Abnormal mammogram or breast examination within the last 9 months suggestive of cancer.
* Abnormal Pap smear or pelvic examination within the last 9 months suggestive of cancer.
* Double-wall endometrial thickness that exceeds 5 mm measured on transvaginal ultrasound.
* Unexplained abnormal uterine bleeding within six months of enrollment.
* Pregnancy or lactating.
* Clinical evidence of active ischemic cardiovascular disease or a history of cardiovascular disease.
* History of deep vein thrombosis or pulmonary embolism requiring anticoagulation.
* Active liver or gallbladder disease.
* Use of medications, herbal or dietary supplements known to possibly be effective for the treatment of hot flashes within three months of enrollment for oral or transdermal drugs, or within 6 months of enrollment for implanted or injected drugs.
* Use of raloxifene or tamoxifen within three months of enrollment.
* Use of another investigational agent within 3 months of enrollment.
* History of multiple or severe food or medicine allergies.
* Any medical or psychiatric condition that, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the trial, including severe illness, plans to move, substance abuse, significant problems, or dementia.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180
Dates: Start 2006-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of hot flashes

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Grady, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota
  - University of Tennessee Health Science Center, Memphis, Tennessee